CLINICAL TRIAL: NCT04814225
Title: A Randomized, Triple-blind, Comparator Controlled, Parallel Clinical Trial to Study the Efficacy and Safety of Three Test Products and Comparator on Muscular Performance in a Healthy, Sedentary Adult Population After the Initiation of a Resistance Training Program
Brief Title: Investigation of the Efficacy and Safety of Three Test Products and Comparator on Muscular Performance After the Initiation of a Resistance Training Program
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roquette Canada, LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 21PMHR
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Muscle Strength
Keywords: pea protein; oat protein; whey protein

STUDY DESIGN:
Intervention Model Description: A randomized, triple-blind, comparator controlled, parallel clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pea Protein Powder (Experimental): Participants will be instructed to mix the IP with 250 mL room temperature water once/day for 12 weeks.
  Interventions: Other: Test Product 1
- Pea & Oat Protein Powder (Experimental): Participants will be instructed to mix the IP with 250 mL room temperature water once/day for 12 weeks.
  Interventions: Other: Test Product 2
- Oat Protein Powder (Experimental): Participants will be instructed to mix the IP with 250 mL room temperature water once/day for 12 weeks.
  Interventions: Other: Test Product 3
- Whey Protein Isolate (Active Comparator): Participants will be instructed to mix the IP with 250 mL room temperature water once/day for 12 weeks.
  Interventions: Other: Comparator

INTERVENTIONS:
Other: Test Product 1 — Pea Protein powder
  Arms: Pea Protein Powder
Other: Test Product 2 — Pea & Oat Protein Powder
  Arms: Pea & Oat Protein Powder
Other: Test Product 3 — Oat Protein Powder
  Arms: Oat Protein Powder
Other: Comparator — Whey Protein Isolate
  Arms: Whey Protein Isolate

SUMMARY:
The objective of this randomized, triple-blind, comparator controlled, parallel clinical trial is to investigate the functional equivalence of three test products compared to whey protein on muscular performance in a healthy, sedentary adult population.

DETAILED DESCRIPTION:
Whey, a by-product of cheese manufacturing, is commonly used as an ingredient in meat products, dairy products, baked goods, snacks, beverages, and infant formula. Its widespread use is due to its advantageous effects on health, economics, and high nutritional value by containing lactose, minerals, vitamins, and soluble proteins. Due to allergies, dietary restrictions and/or personal dietary choices there is a need for an alternative protein source(s), and plant-based protein options are in demand for these reasons. Roquette produces the NUTRALYS® Pea Protein family of ingredients, supplying the widest range of pea protein ingredients to the food industry suitable for use in a plethora of plant-based foods. Few studies have examined the equivalence between pea protein and whey on muscle performance in sedentary adults. The objective of this randomized, triple-blind, comparator controlled, parallel clinical trial is to investigate the functional equivalence of three test products compared to whey protein on muscular performance in a healthy, sedentary adult population.

ELIGIBILITY:
Inclusion Criteria:

1. Males & females between 30 and <60 years of age, inclusive
2. Waist circumference < 102 cm (40 inches) in men and < 88 cm (35 inches) in women
3. Female participant is not of child-bearing potential, defined as females who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least 1 year prior to screening

   Or,

   Females of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
4. Participant having a sedentary lifestyle defined as not engaging in greater than 60 minutes of regular and structured moderate to vigorous exercise per week
5. Self-reported stable body weight for the past 3 months defined as not having gained or lost more than 5 kg of body weight throughout the 3 months prior to baseline
6. Agrees to follow and is able to complete the exercise guidelines for the duration of the study
7. Motivated to comply with exercise guidelines as assessed by the Self-Motivation Questionnaire at screening
8. Agrees to avoid vigorous exercise outside of regular routine for 48 hours prior to and after exercise challenge
9. Agrees to maintain their daily caloric intake
10. Willingness to complete questionnaires, records and diaries associated with the study and to complete all study assessments
11. Willing to refrain from taking NSAID for 24 hours prior to and 72 post study appointments
12. Provided voluntary, written, informed consent to participate in the study
13. Healthy as determined by medical history, laboratory results and electrocardiogram (ECG), as assessed by Qualified Investigator (QI)

Exclusion Criteria:

1. Women who are pregnant, breast feeding, or planning to become pregnant during the study
2. Allergy, sensitivity, or intolerance to the investigational product's active or inactive ingredients. Adheres to a vegan diet
3. Engaged in regular and structured resistance training (≥2x times per week) as assessed by the QI
4. Currently experiencing any medical condition that interferes with the ability to undergo physical strength testing during the study and/or ability to complete exercise guidelines as assessed by the QI
5. Metal implants that may affect the DEXA scan results as assessed on case-by-case basis by the QI
6. Participants who have followed a specific diet (e.g. ketogenic, paleo, etc.) or have had a change of diet within 30 days of baseline as assessed by the QI
7. Current regular use of a protein supplement unless willing to washout (Section 7.3.2)
8. Current use of over-the-counter medications, dietary supplements, foods/drinks for muscle building or function unless willing to washout (Section 7.3.2)
9. Current use of prescribed medications for muscle building or function (see Section 7.3.1)
10. Current use of prescribed steroidal anti-inflammatory medications (see Section 7.3.1), or anti-inflammatory over-the-counter medications or supplements (see Section 7.3.2) unless willing to washout
11. Significant cardiovascular event or revascularization in the past 6 months. Participants with history of cardiovascular event or revascularization will be assessed case by case by the QI. Participants with no significant cardiovascular event on stable medication may be included after assessment by the QI on a case-by-case basis.
12. History of kidney stones will be assessed by the QI on a case-by-case basis
13. Self-reported confirmation of a HIV-, Hepatitis B- or C-positive diagnosis, autoimmune disease or those that are immune compromised
14. Self-reported confirmation of blood/bleeding disorders
15. Alcohol intake >2 standard drinks per day
16. Blood donation 30 days prior to screening, during the study, or a planned donation within 30 days of the last study appointment as assessed by the QI
17. Participation in other pharmaceutical, weight loss/diet, exercise intervention or clinical research studies 30 days prior to enrollment as assessed by the QI
18. Individuals who are unable to give informed consent
19. Any other condition, chronic disease or lifestyle factor, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-04-18 (Actual)

PRIMARY OUTCOMES:
The difference in composite whole-body muscle strength | From baseline to day 84
  The difference in composite whole-body muscle strength, as assessed by the sum of handgrip, elbow flexion and extension and knee flexion and extension strength from baseline to day 84 between IPs 1, 2, 3 and comparator.

SECONDARY OUTCOMES:
The difference in change in handgrip strength | From baseline to days 28, 56 and 84
  The difference in change in muscle strength as assessed by handgrip strength from baseline to days 28, 56 and 84 between IPs 1, 2, 3 and comparator
The difference in change in isometric leg strength | From baseline to days 28, 56 and 84
  The difference in change in muscle strength as assessed by isometric leg strength from baseline to days 28, 56 and 84 between IPs 1, 2, 3 and comparator
The difference in change in upper body strength | From baseline to days 28, 56 and 84
  The difference in change in muscle strength as assessed by upper body strength from baseline to days 28, 56 and 84 between IPs 1, 2, 3 and comparator
The difference in change in weight | From baseline to day 84
  The difference in change in body composition: weight from baseline to day 84 between IPs 1, 2, 3 and comparator
The difference in change in waist circumference | From baseline to day 84
  The difference in change in body composition: waist circumference as assessed by physical measurements from baseline to day 84 between IPs 1, 2, 3 and comparator
The difference in change in android/gynoid fat ratio | From baseline to day 84
  The difference in change in body composition: android/gynoid fat ratio as assessed by DXA from baseline to day 84 between IPs 1, 2, 3 and comparator
The difference in change in fat mass (% or g) | From baseline to day 84
  The difference in change in body composition: fat mass (% or g) as assessed by DXA from baseline to day 84 between IPs 1, 2, 3 and comparator
The difference in change in muscle mass (% or g) | From baseline to day 84
  The difference in change in body composition: muscle mass (% or g) as assessed by DXA from baseline to day 84 between IPs 1, 2, 3 and comparator
The difference in change in endurance performance | From baseline to days 28, 56 and 84
  The difference in change in endurance performance as assessed by Treadmill Walk Test from baseline to days 28, 56 and 84 between IPs 1, 2, 3 and comparator
The difference in change in quality of life | From baseline to days 28, 56 and 84
  The difference in change in quality of life as assessed by RAND SF-36 Quality of Life Questionnaire from baseline to days 28, 56 and 84 between IPs 1, 2, 3 and comparator
The difference in change in blood CRP concentrations | From baseline to days 28, 56 and 84
  The difference in change in blood CRP concentrations from baseline to days 28, 56 and 84 between IPs 1, 2, 3 and comparator
The difference in change in immune function | From screening to day 84
  The difference in change in immune function as assessed by white blood cell (WBC), lymphocyte and neutrophil counts from screening to day 84 between IPs 1, 2, 3 and comparator
The difference in change in product tolerability | From baseline to days 28, 56 and 84
  The difference in change in product tolerability as assessed by Modified Gastrointestinal Symptoms Rating Scale (GSRS) from baseline to days 28, 56 and 84 between IPs 1, 2, 3 and comparator
The difference in product perception | At day 84
  The difference in product perception as assessed by the Product Perception Questionnaire at day 84 between IPs 1, 2, 3 and comparator

OTHER OUTCOMES:
The difference in change in immune function: cytokine response in (TNF)-α | From baseline to days 28, 56 and 84
  The difference in change in immune function as assessed by cytokine response in tumour-necrosis factor (TNF)-α from baseline to days 28, 56 and 84 between IPs 1, 2, 3 and comparator
The difference in change in immune function: cytokine response in IL-6 | From baseline to days 28, 56 and 84
  The difference in change in immune function as assessed by cytokine response in interleukin (IL)-6 from baseline to days 28, 56 and 84 between IPs 1, 2, 3 and comparator
The difference in change in immune function: cytokine response in IL-10 | From baseline to days 28, 56 and 84
  The difference in change in immune function as assessed by cytokine response in IL-10 from baseline to days 28, 56 and 84 between IPs 1, 2, 3 and comparator
Munich ChronoType Questionnaire | At baseline
  The difference in Munich ChronoType Questionnaire (MCTQ) at baseline between IPs 1, 2, 3 and comparator
The difference in change in exercise recovery | At baseline, day 28, 56 and 84
  The difference in change in exercise recovery as assessed by Delayed Onset Muscle Soreness (DOMS) Questionnaire completed 24-, 48-, and 72-hours following the maximum exercise test performed at baseline, day 28, 56 and 84 between IPs 1, 2, 3 and comparator
Incidence of pre-emergent and post-emergent adverse events | From baseline to day 84
  Incidence of pre-emergent and post-emergent adverse events
Blood pressure (BP) | At baseline, day 28, 56 and 84
  Systolic and Diastolic
Heart rate (HR) | At baseline, day 28, 56 and 84
  Heart rate
Aspartate aminotransferase (AST) | At baseline and 84
  Aspartate aminotransferase (AST)
Alanine aminotransferase (ALT) | At baseline and 84
  Alanine aminotransferase (ALT)
Alkaline phosphatase (ALP) | At baseline and 84
  Alkaline phosphatase (ALP)
Total bilirubin | At baseline and 84
  Total bilirubin
Creatinine | At baseline and 84
  Creatinine
Electrolytes (Na, K, Cl) | At baseline and 84
  Electrolytes (Na, K, Cl)
Glucose | At baseline and 84
  Glucose
Estimated glomerular filtration rate (eGFR) | At baseline and 84
  Estimated glomerular filtration rate (eGFR)
Hematology (monocytes, eosinophils, basophils) | At baseline and 84
  Hematology (monocytes, eosinophils, basophils)
Red blood cell (RBC) count | At baseline and 84
  Red blood cell (RBC) count
Hemoglobin | At baseline and 84
  Hemoglobin
Hematocrit | At baseline and 84
  Hematocrit
Platelet count | At baseline and 84
  Platelet count
Mean corpuscular volume (MCV) | At baseline and 84
  RBC indices: mean corpuscular volume (MCV)
Mean corpuscular hemoglobin (MCH) | At baseline and 84
  RBC indices: mean corpuscular hemoglobin (MCH)
Mean corpuscular hemoglobin concentration (MCHC) | At baseline and 84
  RBC indices: mean corpuscular hemoglobin concentration (MCHC)
Red cell distribution width (RDW) | At baseline and 84
  RBC indices: red cell distribution width (RDW)

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science, London, Ontario, Canada